CLINICAL TRIAL: NCT05816187
Title: Study of the Effectiveness and Safety of Supervised Therapeutic Exercise in Cancer Patients With and Without Simultaneous Chemotherapy, Radiotherapy or Hormonal Treatment.
Brief Title: Efficacy and Safety of Supervised Therapeutic Exercise in Cancer Patients With and Without Concurrent Treatment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Hospital Universitario Infanta Leonor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Internal Code 012-23
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Colon Cancer
Keywords: Quality of Life; Therapeutic exercise; Cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised exercise (Experimental): Therapeutic exercise program based on aerobic work, strength-endurance and self-stretching of 6 weeks duration, in addition to a reinforcement of the usual self-care recommendations.
  Interventions: Behavioral: Education program on healthy habits
- Usual care (No Intervention): Subjects receive usual care

INTERVENTIONS:
Behavioral: Education program on healthy habits — 6-week supervised educational program.
  Arms: Supervised exercise

SUMMARY:
OBJECTIVE: To evaluate the effectiveness of a PET scan in oncological patients, with and without simultaneous treatment with chemotherapy, radiotherapy or hormonal therapy, in improving quality of life and the need for supervision by health professionals during its performance after 6 weeks of intervention. DESIGN: Randomized controlled clinical trial, parallel groups with active control group. With randomization blinding, patient assessment and data analysis. STUDY SUBJECTS: 78 patients diagnosed with breast and colon cancer INTERVENTION: two treatment groups: supervised therapeutic exercise and control group. Tho groups will be supervised in performing PET for a period of 6 weeks and the other group will receive the usual care. Patients will be followed for 1 year, with five blinded assessments: at baseline, after 6 weeks of intervention, 3, 6 and 12 months after baseline. MEASUREMENTS: Main: Quality of life assessed with questionnaire measured with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC QLQ-30). Measured pre-post intervention, 3, 6 and 12 months. Secondary: Cancer-related fatigue assessed with the Functional Assessment of scale Chronic Illness Therapy - Fatigue (FACIT-F). Measured pre-post intervention, 3, 6 and 12 months. Functional capacity measured with the 6-minute walk test. Pre-post intervention measurement, 3, 6 and 12 months. Strength assessment measured with manual hydraulic dynamometer and 5 repetitions of the sit-to-stand test. Pre-post intervention measurement, 3, 6 and 12 months.

DETAILED DESCRIPTION:
OBJECTIVE: To evaluate the effectiveness of a PET scan in oncological patients, with and without simultaneous treatment with chemotherapy, radiotherapy or hormonal therapy, in improving quality of life and the need for supervision by health professionals during its performance after 6 weeks of intervention. DESIGN: Randomized controlled clinical trial. With randomization blinding, patient assessment and data analysis. STUDY SUBJECTS: 78 patients diagnosed with breast and colon cancer . INTERVENTION: two treatment groups: supervised therapeutic exercise group and control group. Intevention group will be supervised in performing PET for a period of 6 weeks and the other group will receive the usual care. Patients will be followed for 1 year, with five blinded assessments: at baseline, after 6 weeks of intervention, 3, 6 and 12 months after baseline. MEASUREMENTS: Main: Quality of life assessed with questionnaire measured with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC QLQ-30). Measured pre-post intervention, 3, 6 and 12 months. Secondary: Cancer-related fatigue assessed with the Functional Assessment of scale Chronic Illness Therapy - Fatigue (FACIT-F). Measured pre-post intervention, 3, 6 and 12 months. Functional capacity measured with the 6-minute walk test. Pre-post intervention measurement, 3, 6 and 12 months. Strength assessment measured with manual hydraulic dynamometer and 5 repetitions of the sit-to-stand test. Pre-post intervention measurement, 3, 6 and 12 months.COST

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years.
* Oncological stage I, II or III.
* Completed adjuvant treatment between 3 months to 2 years. ECOG 1-2.
* Sign informed consent

Exclusion Criteria:

* Inability to read, understand and complete questionnaires, read and understand a brochure explanatory, understand and follow verbal orders (example; illiteracy, dementia or blindness).
* Musculoskeletal disorders that prevent the exercise of the exercise bike, elliptical, march tape.
* Important neurological disorders that involve impaired balance, coordination, ataxia.
* Sporting activity at moderate intensity exceeding 150mnts / week.
* Symptomatic anemia.
* Fecal incontinence
* Patient with a digestive ostomy.
* Decompensated heart disease,
* Uncontrolled hypertension
* Heart failure.
* Musculoskeletal pathology (except for upper limb pathology in cancer patients of mom)
* Cardio-respiratory pathology that limits physical activity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Changes in Health Related Quality of Life: EORTC QLQ-30 | Basal, 1.5, 3, 6, 12 months follow up
  (EORTC QLQ-30). The QLQ-C30 questionnaire is a specific questionnaire for cancer, it is composed of 30 questions or items that assess the quality of life in relation to physical, emotional, social aspects and in general the level of functionality of patients diagnosed with cancer. The QLQ-C30 questionnaire is assigned values between 1 and 4 (1: not at all, 2: a little, 3: a lot, 4: a lot) according to the patient's responses to the item, only in items 29 and 30 are assessed with score from 1 to 7 (1: bad, 7: excellent). The scores obtained are standardized and a score between 0 and 100 is obtained, 0 being the worst possible and 100 the best.

SECONDARY OUTCOMES:
Fatigue measurement with FACIT-F | 1.5, 3, 6, 12 months follow up
  Fatigue measurement with FACIT-F (Functional Assessment of Chronic Illness Therapy-Fatigue) questionaire.
  The FACIT-F 13-item scale is designed on a 5-point Likert scale (0 = nothing; 1 = little; 2 = something; 3 = a lot; 4 = very much). The FACIT-F scale is designed so that a high score is good, the possible score is 0 to 52, 0 being the worst possible and 52 the best.
Functional capacity | Basal, 1.5, 3, 6, 12 months follow up
  The 6-minute walk test consists of measuring the maximum distance that the patient is able to walk in 6 minutes, on a tour short in a hallway, simultaneously assessing heart rate, oxygen saturation and degree of dyspnea. Usually healthy people can walk between 400 and 700 meters in 6 minutes, depending on age, height and sex
Force with manual hydraulic dynamometer. | Basal, 1.5, 3, 6, 12 months follow up
  Valuation of the measured force with manual hydraulic dynamometer . The prehensile force exerted during 5 seconds will be measured, it will be done 3 times and the average will be taken.
The five Times Sit to Stand Test (5x Sit-To-Stand Test) | Basal, 1.5, 3, 6, 12 months follow up
  Valuation of the functional lower extremity strength with the The five Times Sit to Stand Test (5x Sit-To-Stand Test), The 5XSST scoring is based on the amount of time (to the nearest decimal in seconds) a patient is able to transfer from a seated to a standing position and back to sitting five times. The equipment need in performing 5XSST test includes: Stopwatch and standard height chair with straight back (43-45 cm, 17-18 inches high). Then the instruction is given by asking the test taker to sit on the chair by resting their back. Also, the test taker is instructed to fold their arms across their chest. Then the test taker should be instructed to do sit-to-stand five times, as quickly as possible, at the count of go and without their back or leg resting on the chair between the interval of repetition.
  The lower the time to complete the test the better the outcome of the test.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Infanta Leonor, Madrid, Spain